CLINICAL TRIAL: NCT00726570
Title: Effects of Sequential Compression Devices on Coagulation Parameters Assessed by TEG® in Patients Undergoing Major Abdominal Surgery
Brief Title: Alterations of Blood Clotting With the Use of Sequential Compression Devices on the Lower Limbs
Acronym: TEGLeg
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to reach the expected enrollment rates by the end of 2010
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Guido Fanelli, MD, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ICU-ICU-01
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Coagulation, Blood; Compression Devices, Intermittent Pneumatic; Postoperative Complications; Thrombelastography
Keywords: Disorders, Blood coagulation; Deep Vein Thrombosis; Perioperative Care; Digestive System Surgical Procedures
MeSH Terms: conditions — Thrombosis; Postoperative Complications; Blood Coagulation Disorders; Venous Thrombosis | interventions — Dalteparin; Heparin, Low-Molecular-Weight; Heparin; Anticoagulants; Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCD + LMWH (Experimental): This group will receive sequential compression device therapy to the lower limbs from their ICU admission until the morning after surgery.
  Interventions: Device: Sequential compression device therapy; Drug: Dalteparin; Procedure: TEG
- LMWH only (Active Comparator): Patients in this group will receive only standard LMWH therapy during their ICU stay.
  Interventions: Drug: Dalteparin; Procedure: TEG

INTERVENTIONS:
Device: Sequential compression device therapy — Pneumatic stockings will be applied to patients.
  Pressures ranging from 12 to 40 mmHg will be applied at different levels of the lower limb for 40-second cycles at 2-minute intervals. Therapy will continue until the morning after surgery.
  Other Names: SCD EXPRESS; Foot pump
  Arms: SCD + LMWH
Drug: Dalteparin — * 2500 UI qd if ≤ 50 kg body weight
  * 5000 UI qd if > 50 kg
  Other Names: low molecular weight heparin; Fragmin; heparin; thromboprophylaxis; anticoagulant; LMWH
Procedure: TEG — A 2-ml blood sample will be used for each exam. A full analysis will be run both with and without heparinase at each time point.
  TEG analyses will be run at:
  * Patient admission (before SCD start)
  * 40-60 min after admission
  * Morning after surgery
  Other Names: thrombelastography; TEG®; thrombelastogram

SUMMARY:
This study aims to assess possible alteration in coagulation (blood clotting) following treatment with sequential compression devices (SCD) plus low-molecular weight heparin (LMWH) as opposed to LMWH alone.

The investigators will examine coagulation in the early postoperative period of patients undergoing major abdominal surgery during their stay in our Intensive Care Unit.

In addition to common laboratory tests, the investigators will examine coagulation using TEG®, a device which allows a semi-quantitative examination of all phases of coagulation.

DETAILED DESCRIPTION:
Low molecular weight heparins (LMWH) are routinely used in perioperative prophylaxis of thromboembolic complications [(chiefly deep vein thrombosis (DVT)]. LMWHs have been proved to be safe and equipotent or superior when compared with unfractionated heparin.

Sequential compressing devices (SCD) are relatively novel pneumatic stockings with several air chambers. A computerized pump applies a gradient of pressure which decreases from the foot cranially. Pressure is also applied intermittently according to predetermined schedules. This devices are being employed for DVT prophylaxis in patients for whom anticoagulation therapy is contraindicated, or in those who have a low risk of DVT. They have also been employed to complement anticoagulant therapy in patients at high risk of DVT, such as those undergoing orthopedic surgery (Fordyce, 1992; Handoll, 2002; Warwick, 2002; Pitto, 2004).

The mechanism of action of SCD seems to be primarily mechanical, through a displacement of a column of blood through the venous system and towards the heart; they act as a surrogate of the muscular pump in immobilized patients (Killewich, 1995).

There is also some evidence that SCD activity may influence the coagulation/fibrinolysis system towards hypocoagulability (Dai, 2000; Kohro, 2003); Kohro and colleagues have also hypothesized that the shear forces generated by SCD may alter platelet adhesion by a direct effect on platelets and/or by increasing the release of factors from the venous endothelium (Kohro, 2005).

The investigators aim to assess the effects on coagulation when SCD are applied to patients at high risk of DVT in addition to standard LMWH therapy.The investigators chose to study a population in whom SCD may be useful in reducing the incidence of DVT, such as patients undergoing postoperative monitoring in the intensive care unit (ICU) after major abdominal surgery for cancer.

In addition to standard laboratory tests, the investigators will use thrombelastography (TEG®) to assess all phases of coagulation. A TEG parameter, maximum amplitude (MA), has been linked to an increase of thrombotic complications in a postoperative population (McCrath, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Elective major abdominal surgery for neoplasm
* Planned admission to postsurgical ICU due to the patient's meeting one or more of the following:

  * ASA Physical Status Class 4
  * Surgery of modified Johns-Hopkins class ≥IV
  * ASA 3 with modified Johns-Hopkins class 3 surgery
  * Expected duration of surgery ≥8 h

Exclusion Criteria:

* History of coagulation abnormalities, either congenital or acquired
* Ongoing treatment with anticoagulants/antiplatelet agents other than LMWH or hormones
* Massive edema of the legs
* Severe peripheral arteriopathy or neuropathy
* Malformations or recent surgery/trauma to the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the area under the curve of maximum amplitude (MA) TEG value over time | 24 hours from application of SCD

SECONDARY OUTCOMES:
Reduction in the area under the curve of the r time TEG value over time | 24 h after application of SCD
Reduction in the area under the curve of the alpha angle TEG value over time | 24 h after application of SCD
Incidence of hypotension (mean arterial pressure ≤60 mmHg) | ≤24 h after application of SCD

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Study Chair — University of Parma; Maria Barbagallo, MD, Principal Investigator — UO II Anestesia e Rianimazione, Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- University Hospital / Azienda Ospedaliero-Universitaria, Parma, PR, Italy

REFERENCES:
- [Background] Fordyce MJ, Ling RS. A venous foot pump reduces thrombosis after total hip replacement. J Bone Joint Surg Br. 1992 Jan;74(1):45-9. doi: 10.1302/0301-620X.74B1.1732264.
- [Background] Handoll HH, Farrar MJ, McBirnie J, Tytherleigh-Strong G, Milne AA, Gillespie WJ. Heparin, low molecular weight heparin and physical methods for preventing deep vein thrombosis and pulmonary embolism following surgery for hip fractures. Cochrane Database Syst Rev. 2002;(4):CD000305. doi: 10.1002/14651858.CD000305. PMID 12519540
- [Background] Warwick D, Harrison J, Whitehouse S, Mitchelmore A, Thornton M. A randomised comparison of a foot pump and low-molecular-weight heparin in the prevention of deep-vein thrombosis after total knee replacement. J Bone Joint Surg Br. 2002 Apr;84(3):344-50. doi: 10.1302/0301-620x.84b3.12372. PMID 12002490
- [Background] Pitto RP, Hamer H, Heiss-Dunlop W, Kuehle J. Mechanical prophylaxis of deep-vein thrombosis after total hip replacement a randomised clinical trial. J Bone Joint Surg Br. 2004 Jul;86(5):639-42. doi: 10.1302/0301-620x.86b5.14763. PMID 15274256
- [Background] Killewich LA, Sandager GP, Nguyen AH, Lilly MP, Flinn WR. Venous hemodynamics during impulse foot pumping. J Vasc Surg. 1995 Nov;22(5):598-605. doi: 10.1016/s0741-5214(95)70046-3. PMID 7494362
- [Background] Dai G, Tsukurov O, Orkin RW, Abbott WM, Kamm RD, Gertler JP. An in vitro cell culture system to study the influence of external pneumatic compression on endothelial function. J Vasc Surg. 2000 Nov;32(5):977-87. doi: 10.1067/mva.2000.110357. PMID 11054230
- [Background] Kohro S, Yamakage M, Takahashi T, Ota K, Kondo M, Namiki A. Effects of intermittent pneumatic foot compression on blood coagulability and fibrinolysis assessed by a whole blood viscometer Sonoclot. J Anesth. 2003;17(3):208-10. doi: 10.1007/s00540-003-0180-x. No abstract available. PMID 12911214
- [Background] Kohro S, Yamakage M, Sato K, Sato JI, Namiki A. Intermittent pneumatic foot compression can activate blood fibrinolysis without changes in blood coagulability and platelet activation. Acta Anaesthesiol Scand. 2005 May;49(5):660-4. doi: 10.1111/j.1399-6576.2005.00661.x. PMID 15836680
- [Background] McCrath DJ, Cerboni E, Frumento RJ, Hirsh AL, Bennett-Guerrero E. Thromboelastography maximum amplitude predicts postoperative thrombotic complications including myocardial infarction. Anesth Analg. 2005 Jun;100(6):1576-1583. doi: 10.1213/01.ANE.0000155290.86795.12. PMID 15920177